CLINICAL TRIAL: NCT04846998
Title: A Randomized, Open-label, Three-treatment, Six-sequence, Three-period, Crossover Clinical Study to Compare the Pharmacokinetic Characteristics Between Twice Daily Administration of BR9003A and Once Daily Administration of BR9003 in Healthy Adult Subjects
Brief Title: A Study to Compare the Pharmacokinetics of BR9003A and BR9003 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-VRNS-CT-102
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 1: A-B-C
  Interventions: Drug: BR9003; Drug: BR9003A
- Sequence 2 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 2: A-C-B
  Interventions: Drug: BR9003; Drug: BR9003A
- Sequence 3 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 3: B-A-C
  Interventions: Drug: BR9003; Drug: BR9003A
- Sequence 4 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 4: B-C-A
  Interventions: Drug: BR9003; Drug: BR9003A
- Sequence 5 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 5: C-A-B
  Interventions: Drug: BR9003; Drug: BR9003A
- Sequence 6 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 6: C-B-A
  Interventions: Drug: BR9003; Drug: BR9003A

INTERVENTIONS:
Drug: BR9003 — Treatment group B:
  Once-daily oral administration of one BR9003 2mg tablet in the fasting state.
  Treatment group C:
  Once-daily oral administration of one BR9003 2mg tablet after a meal(high-fat meal) 30 minutes before the scheduled time of administration and finishing it.
Drug: BR9003A — Treatment group A:
  Twice-daily oral administration of one BR9003A 1mg tablet in the fasting state

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of oral administration of BR9003 compared with BR9003A in healthy adult subjects

DETAILED DESCRIPTION:
A total of 24 subjects will be randomized into 6 sequence groups. The Investigational Products wil be according to the treatment group (A,B,C) assigned to each sequence group in Period 1, Period 2 and Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years at screening
2. Those who weigh at least 50 kg at the time of screening and have a calculated body mass index (BMI) within the range of 18.0 to 29.0 kg/m2
3. Determined to be eligible as subjects through physical examination and interview conducted in accordance with this protocol. In other words, those who have no congenital or chronic diseases and have no abnormal symptoms or findings based on medical examination results within the last 3 years
4. Determined to be eligible as subjects as a result of clinical laboratory tests and electrocardiography performed according to this protocol
5. Voluntarily decide to participate in the study and provide written consent to follow the study directions after listening to and fully understanding the detailed explanation on this study

Exclusion Criteria:

1. Those who have clinically significant diseases or a history of the diseases associated with the cardiovascular system, respiratory system, liver, kidney, nervous system, endocrine system, blood/tumor, psychiatric diseases, or urinary system
2. Those who have hypersensitivity reactions or a history of clinically significant hypersensitivity reactions to drugs containing varenicline, or drugs containing the same class ingredients, or other drugs
3. Those with clinically significant hypotension (systolic blood pressure ≤ 90mmHg) or hypertension (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 95mmHg) at the time of screening
4. Those with a history of gastrointestinal diseases (e.g., Crohn's disease, ulcer, etc.) or gastrointestinal surgery (however, simple appendectomy or hernia repair are excluded) that may affect the absorption of drugs
5. Any of the following results in the screening tests

   * AST or ALT > 2 times the upper limit of the normal range
   * Total bilirubin > 2.0 mg/dL
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
6. Those who continue to drink alcohol (>21 units/week; 1 unit = 10 g = 12.5 mL of pure alcohol), or are unable to abstain from drinking during the clinical study period
7. Those who continue to smoke (>10 cigarettes/day) or cannot stop smoking during hospitalization during the clinical trial period
8. Those who have participated in another clinical trial or bioequivalence test (the last day of administration of the investigational product or bioequivalence test drug) within 6 months prior to the first administration date
9. Those who have donated whole blood within 60 days prior to the first day of administration or donated blood components (apheresis) within 30 days prior to the first day of administration or who have received a blood transfusion within 30 days
10. Those who took any prescription drugs or herbal medicines within 14 days prior to the first day of administration or any over-the-counter (OTC) drugs within 7 days prior to the first day of administration (however, if other conditions are appropriate according to the judgment of the investigator, they may participate in the clinical trial.)
11. Those who took drugs inducing and inhibiting drug-metabolizing enzymes, such as barbital, within 30 days prior to the study initiation
12. Those who have been on a diet (especially grapefruit juice or its products) that may affect the absorption, distribution, metabolism, and excretion of the drug within 7 days prior to the first day of administration
13. Pregnant woman, potentially pregnant woman, or breast-feeding woman
14. Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy using a medically acceptable methods of contraception* throughout the entire period from the date of the first administration of the investigational product to the end of the clinical trial
15. Those who are unwilling or unable to comply with the dietary and lifestyle guidelines required for the clinical trial
16. Those who have clinically significant abnormalities in the results of other clinical laboratory tests or who have been determined by the investigator to be ineligible to participate in the clinical trial due to other reasons (e.g., non-compliance with instructions, uncooperative attitude, etc.)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-72 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time t of BR9003 and BR9003A
Cmax | 0-72 hours after administration
  Maximum concentration of drug in plasma of BR9003 and BR9003A

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No